CLINICAL TRIAL: NCT06427655
Title: Benefit of the SALAD Technique on CPR Quality During Intubation in Contaminated Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20220903R
Record Dates: First submitted 2024-05-12; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Airway Aspiration; Cardiopulmonary Arrest
Keywords: airway decontamination; suction assisted; resuscitation; cardiopulmonary resuscitation quality
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two groups. One group utilizing the SALAD technique and the other employing intermittent suction during intubation on a manikin.
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent suction (No Intervention): intermittent suction during intubation
- SALAD (Experimental): SALAD suction during intubation
  Interventions: Device: SALAD intubation

INTERVENTIONS:
Device: SALAD intubation — SALAD suction during intubation
  Arms: SALAD

SUMMARY:
Management of airways in contaminated environments can compromise the quality of cardiopulmonary resuscitation (CPR). This study examined the effectiveness of SALAD (Suction Assisted Laryngoscopy Airway Decontamination) compared to intermittent suction in maintaining CPR quality during intubation in a simulated scenario of regurgitation. Following 2.5 hours of training in the SALAD technique, 36 emergency medicaltechnician-paramedics (EMT-Ps) were randomly assigned in equal numbers to two groups: one utilizing the SALAD technique and the other employing intermittent suction during intubation on a manikin. The manikin simulates regurgitation of gastric contents into the oropharynx during CPR. Primary outcomes assessed were CPR quality metrics, such as chest compression rate, depth, and interruption. Secondary outcomes included the success rate and time of intubation.

DETAILED DESCRIPTION:
The study was conducted in March 2024. Participants were emergency medical technician-paramedics (EMT-Ps) employed by fire departments across Taiwan, recruited on a nationwide basis. All participants provided signed informed consent forms. 36 EMT-Ps are involved in this study.

Simulation setup :

The CPR-induced regurgitation model was adapted from an Airway Larry Airway Management Trainer Torso (Nasco, Fort Atkinson, WI, USA) to simulate oropharyngeal regurgitation during CPR. To emulate the stomach, a manual pump was attached at the base of the manikin's torso. A transparent vinyl tube connected the manikin's esophagus to the pump's outlet port. A HQCPR device was used for CPR quality record.

Training program The 36 participants received 2.5 hours of SALAD training. The training included 5 rounds of intubation teaching and practice. The first two rounds of training involve using the SALAD technique with the video laryngoscope, while the third round used the C-MAC S video laryngoscope as a direct laryngoscope for practice. Technique adjustments can be made during the initial three rounds through monitoring with the video system. The fourth round will involve intubation using a direct laryngoscope with a size 3 Macintosh blade on the SALAD Simulator. The final round involved intubation on the CPR-induced regurgitation model, using a direct laryngoscope and employing the SALAD technique for intubation during chest compressions.

Simulation protocol After completing 2.5 hours of training, participants were randomly assigned to one of two groups for suction techniques: SALAD or intermittent suction. Randomization was conducted using the simple randomization method with a random number table. Participants assigned to the same suction technique group formed a resuscitation team, taking on roles as the airway manager, first chest compressor, or second chest compressor. Each participant rotated through these three roles during three simulation sessions.In each simulation, the airway manager was responsible for BVM ventilation and intubation. The first and second chest compressors performed chest compressions alternately, once every five CPR cycles, adhering to a 30:2 compression-to- ventilation ratio. The initial 30 chest compressions were followed by two ventilations, and suction was not performed during this phase, even if regurgitation was present. This was intended to simulate a scenario where the oral cavity was filled with regurgitant material during intubation, maintaining consistency across participants. After the first two ventilations, intubation could proceed while the team continued chest compressions. The airway manager could request a temporary reduction, lightening, or even cessation of chest compressions to facilitate intubation, or to continue up to 60 compressions without interruption if necessary. If the intubation attempt was unsuccessful, the airway manager had to administer two BVM ventilations before attempting intubation again. Depending on the group assignment, either SALAD or intermittent suction techniques were employed to assist in airway decontamination. After intubation, the airway manager assessed lung expansion using the BVM to verify successful intubation. A failed intubation was defined as any esophageal intubation or three unsuccessful intubation attempts. Each simulation concluded following either a successful or failed intubation.

Measurement The primary outcomes were CPR quality metrics, including chest compression rate, chest compression depth, and time of interruption. The secondary outcomes were the intubation success rate and intubation time. The rate and depth of the first 30 chest compressions (pre-intubation period) were measured. After the initial 30 compressions, interruptions for ventilation or airway management, as well as the quality of chest compressions during intubation, were also measured (intubation period). An intubation attempt was defined as the insertion of the laryngoscope blade into the mouth and its subsequent withdrawal during an unsuccessful attempt, or as the insertion of the laryngoscope blade followed by confirmation from the airway manager that the tube was inserted. Intubation time was defined as the period between the start and the end of an intubation attempt. Two video cameras were set up to record the entire simulation process. Two observers reviewed the video records independently to identify any intubation attempts. Disagreements were resolved by reaching a mutual consensus.

The HQCPR application on an Android device recorded chest compression depth, rate, and interruptions (defined as no chest compression for more than 1 second).

The data from both the video recordings and the HQCPR application were used in subsequent analyses.

Statistical analysis The characteristics of EMT-Ps were described using frequency and percentage for categorical variables, while mean values with standard deviation (SD) were used for continuous variables. Continuous data were compared using the independent t-test between the SALAD and intermittent suction groups, while categorical data were compared using the Fisher's exact test or the Chi-Squared test between these two groups. CPR quality metrics and intubation time were summarized using mean values with 95% confidence intervals (CI). Compression depth greater than or equal to 5 cm, first-pass intubation success, and esophageal intubation were presented as frequency and percentage. Continuous data were compared using the independent t test between the SALAD and intermittent suction groups, while categorical data were compared using Fisher's exact test between these two groups. CPR quality metrics between the pre-intubation period and the intubation period were analyzed using the paired t test in both the SALAD and intermittent suction groups. A two- tailed p-value of less than 0.05 indicated statistical significance. All data analyses and sample size determination were performed using MedCalc Statistical Software version 22.023 (MedCalc Software, Ostend, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* emergency medical technician-paramedics experienced in advanced airway management and CPR

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
chest compression fraction | 3 hour
  the proportion of time spent performing chest compressions during arrest

SECONDARY OUTCOMES:
success rate of intubation | 3 hour
  the rate of successful intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Shinkong Wu-Ho-Su memorial hospital, Taipei, Shih-Lin, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simons RW, Rea TD, Becker LJ, Eisenberg MS. The incidence and significance of emesis associated with out-of-hospital cardiac arrest. Resuscitation. 2007 Sep;74(3):427-31. doi: 10.1016/j.resuscitation.2007.01.038. Epub 2007 Apr 11. PMID 17433526
- [Background] Benger JR, Kirby K, Black S, Brett SJ, Clout M, Lazaroo MJ, Nolan JP, Reeves BC, Robinson M, Scott LJ, Smartt H, South A, Stokes EA, Taylor J, Thomas M, Voss S, Wordsworth S, Rogers CA. Effect of a Strategy of a Supraglottic Airway Device vs Tracheal Intubation During Out-of-Hospital Cardiac Arrest on Functional Outcome: The AIRWAYS-2 Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):779-791. doi: 10.1001/jama.2018.11597. PMID 30167701
- [Background] Wang HE, Simeone SJ, Weaver MD, Callaway CW. Interruptions in cardiopulmonary resuscitation from paramedic endotracheal intubation. Ann Emerg Med. 2009 Nov;54(5):645-652.e1. doi: 10.1016/j.annemergmed.2009.05.024. Epub 2009 Jul 2. PMID 19573949
- [Background] Ruetzler K, Gruber C, Nabecker S, Wohlfarth P, Priemayr A, Frass M, Kimberger O, Sessler DI, Roessler B. Hands-off time during insertion of six airway devices during cardiopulmonary resuscitation: a randomised manikin trial. Resuscitation. 2011 Aug;82(8):1060-3. doi: 10.1016/j.resuscitation.2011.03.027. Epub 2011 Apr 6. PMID 21514986
- [Background] Wang HE, Jaureguibeitia X, Aramendi E, Jarvis JL, Carlson JN, Irusta U, Alonso E, Aufderheide T, Schmicker RH, Hansen ML, Huebinger RM, Colella MR, Gordon R, Suchting R, Idris AH. Airway strategy and chest compression quality in the Pragmatic Airway Resuscitation Trial. Resuscitation. 2021 May;162:93-98. doi: 10.1016/j.resuscitation.2021.01.043. Epub 2021 Feb 11. PMID 33582258
- [Background] Wang HE, Schmicker RH, Daya MR, Stephens SW, Idris AH, Carlson JN, Colella MR, Herren H, Hansen M, Richmond NJ, Puyana JCJ, Aufderheide TP, Gray RE, Gray PC, Verkest M, Owens PC, Brienza AM, Sternig KJ, May SJ, Sopko GR, Weisfeldt ML, Nichol G. Effect of a Strategy of Initial Laryngeal Tube Insertion vs Endotracheal Intubation on 72-Hour Survival in Adults With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):769-778. doi: 10.1001/jama.2018.7044. PMID 30167699
- [Background] Piegeler T, Roessler B, Goliasch G, Fischer H, Schlaepfer M, Lang S, Ruetzler K. Evaluation of six different airway devices regarding regurgitation and pulmonary aspiration during cardio-pulmonary resuscitation (CPR) - A human cadaver pilot study. Resuscitation. 2016 May;102:70-4. doi: 10.1016/j.resuscitation.2016.02.017. Epub 2016 Feb 26. PMID 26921473
- [Background] Lin LW, DuCanto J, Hsu CY, Su YC, Huang CC, Hung SW. Compromised cardiopulmonary resuscitation quality due to regurgitation during endotracheal intubation: a randomised crossover manikin simulation study. BMC Emerg Med. 2022 Jul 9;22(1):124. doi: 10.1186/s12873-022-00662-0. PMID 35810275
- [Background] DuCanto J, Serrano KD, Thompson RJ. Novel Airway Training Tool that Simulates Vomiting: Suction-Assisted Laryngoscopy Assisted Decontamination (SALAD) System. West J Emerg Med. 2017 Jan;18(1):117-120. doi: 10.5811/westjem.2016.9.30891. Epub 2016 Nov 8. PMID 28116021
- [Background] Lin LW, Huang CC, Ong JR, Chong CF, Wu NY, Hung SW. The suction-assisted laryngoscopy assisted decontamination technique toward successful intubation during massive vomiting simulation: A pilot before-after study. Medicine (Baltimore). 2019 Nov;98(46):e17898. doi: 10.1097/MD.0000000000017898. PMID 31725637
- [Background] Pilbery R, Teare MD. Soiled airway tracheal intubation and the effectiveness of decontamination by paramedics (SATIATED): a randomised controlled manikin study. Br Paramed J. 2019 Jun 1;4(1):14-21. doi: 10.29045/14784726.2019.06.4.1.14. PMID 33328824
- [Background] Fiore MP, Marmer SL, Steuerwald MT, Thompson RJ, Galgon RE. Three Airway Management Techniques for Airway Decontamination in Massive Emesis: A Manikin Study. West J Emerg Med. 2019 Aug 6;20(5):784-790. doi: 10.5811/westjem.2019.6.42222. PMID 31539335
- [Background] Kleinman ME, Brennan EE, Goldberger ZD, Swor RA, Terry M, Bobrow BJ, Gazmuri RJ, Travers AH, Rea T. Part 5: Adult Basic Life Support and Cardiopulmonary Resuscitation Quality: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S414-35. doi: 10.1161/CIR.0000000000000259. No abstract available. PMID 26472993
- [Background] Agostinucci JM, Weisslinger L, Marzouk N, Zouaghi H, Ekpe K, Genthillomme A, Adnet F, Guenin A, Reuter PG, Lapostolle F. Relation between chest compression rate and depth: the ENFONCE Study. Eur J Emerg Med. 2021 Oct 1;28(5):352-354. doi: 10.1097/MEJ.0000000000000802. PMID 33758145
- [Background] McAlister O, Harvey A, Currie H, McCartney B, Adgey J, Owens P, Idris A. Temporal analysis of continuous chest compression rate and depth performed by firefighters during out of hospital cardiac arrest. Resuscitation. 2023 Apr;185:109738. doi: 10.1016/j.resuscitation.2023.109738. Epub 2023 Feb 16. PMID 36806652
- [Background] Stiell IG, Brown SP, Nichol G, Cheskes S, Vaillancourt C, Callaway CW, Morrison LJ, Christenson J, Aufderheide TP, Davis DP, Free C, Hostler D, Stouffer JA, Idris AH; Resuscitation Outcomes Consortium Investigators. What is the optimal chest compression depth during out-of-hospital cardiac arrest resuscitation of adult patients? Circulation. 2014 Nov 25;130(22):1962-70. doi: 10.1161/CIRCULATIONAHA.114.008671. Epub 2014 Sep 24. PMID 25252721
- [Background] Voss S, Rhys M, Coates D, Greenwood R, Nolan JP, Thomas M, Benger J. How do paramedics manage the airway during out of hospital cardiac arrest? Resuscitation. 2014 Dec;85(12):1662-6. doi: 10.1016/j.resuscitation.2014.09.008. Epub 2014 Sep 26. PMID 25260723
- [Background] Deakin CD, Nolan JP, Ji C, Fothergill RT, Quinn T, Rosser A, Lall R, Perkins GD. The effect of airway management on CPR quality in the PARAMEDIC2 randomised controlled trial. Resuscitation. 2021 Jan;158:8-13. doi: 10.1016/j.resuscitation.2020.11.005. Epub 2020 Nov 12. PMID 33189805
- [Background] Donoghue A, Hsieh TC, Nishisaki A, Myers S. Tracheal intubation during pediatric cardiopulmonary resuscitation: A videography-based assessment in an emergency department resuscitation room. Resuscitation. 2016 Feb;99:38-43. doi: 10.1016/j.resuscitation.2015.11.019. Epub 2015 Dec 17. PMID 26703462
- [Background] Robinson AE, Driver BE, Prekker ME, Reardon RF, Horton G, Stang JL, Collins JD, Carlson JN. First attempt success with continued versus paused chest compressions during cardiac arrest in the emergency department. Resuscitation. 2023 May;186:109726. doi: 10.1016/j.resuscitation.2023.109726. Epub 2023 Feb 9. PMID 36764570
- [Background] Murphy DL, Bulger NE, Harrington BM, Skerchak JA, Counts CR, Latimer AJ, Yang BY, Maynard C, Rea TD, Sayre MR. Fewer tracheal intubation attempts are associated with improved neurologically intact survival following out-of-hospital cardiac arrest. Resuscitation. 2021 Oct;167:289-296. doi: 10.1016/j.resuscitation.2021.07.001. Epub 2021 Jul 14. PMID 34271128
- [Background] Jost D, Minh PD, Galinou N, Alhanati L, Dumas F, Lemoine F, Tourtier J-P. What is the incidence of regurgitation during an out-of-hospital cardiac arrest? Observational study Resuscitation. 2015;96:70.
- [Background] Ko S, Wong OF, Wong CHK, Ma HM, Lit CHA. A pilot study on using Suction-Assisted Laryngoscopy Airway Decontamination techniques to assist endotracheal intubation by GlideScope® in a manikin simulating massive hematemesis. Hong Kong Journal of Emergency Medicine. 2021;28(5):305-313.
- [Background] Choi I, Choi YW, Han SH, Lee JH. Successful endotracheal intubation using suction- assisted laryngoscopy assisted decontamination technique and a head-down tilt position during massive regurgitation. Soonchunhyang Med Sci. 2020; 26 ( 2 ):75-9.
- [Background] Frantz E, Sarani N, Pirotte A, Jackson BS. Woman in respiratory distress. J Am Coll Emerg Physicians Open. 2021 Jan 14;2(1):e12344. doi: 10.1002/emp2.12344. eCollection 2021 Feb. No abstract available. PMID 33490996
- [Background] Vittinghus, S., Thomsen, J.E., Harpsø, M. Bo Løfgren. Does the age of medical emergency technicians influence the quality of chest compressions. Scand J Trauma Resusc Emerg Med. 2015;23 (Suppl 1): A9
- See also: Related Info — https://www.anesthesiologynews.com/Review-Articles/Article/07-23/Airway-Contamination-To-Stop-or-Continue-CPR-During-Intubation-Attempts/70740?ses=ogst